CLINICAL TRIAL: NCT05743829
Title: Atrial Fibrillation Driver Study - Pilot Project
Brief Title: Atrial Fibrillation Driver Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CAR0630
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation; Fibrosis Myocardial
Keywords: AF; Fibrosis
MeSH Terms: conditions — Atrial Fibrillation; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In all cases tissue that is surplus to the clinical requirement will be obtained if available. This tissue will be either processed for histological analyses (including embedding for immunohistochemistry, in situ hybridisation, electron microscopy), flash frozen in liquid nitrogen for assays including collagen cross-linking, or cultured in vitro and stimulated with relevant stimuli. These analyses may be complemented by additional assays (including but not limited to) for genome sequencing, miRNA and RNA sequencing, culture, RT-PCR, flow cytometry and immunocytochemistry. Cells established in culture will also be stored in liquid nitrogen for experimental investigations at later dates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiac Surgery: Patients undergoing cardiac surgery - left atrial appendage excision
  Interventions: Procedure: Tissue excision as part of routine clinical care
- Thoracic Surgery: Patients undergoing lung resection - ostial pulmonary vein tissue
  Interventions: Procedure: Tissue excision as part of routine clinical care

INTERVENTIONS:
Procedure: Tissue excision as part of routine clinical care — Tissue excision

SUMMARY:
Atrial Fibrillation (AF) is an abnormal rhythm of the heart which is increasingly common and can be associated with serious consequences. We know that AF is associated with an increase in the scarring of the heart, the left atrium and it is thought that this scarring may be one of the drivers for this abnormal heart rhythm. The nature of this scarring in humans has been subject to limited study and generally only by indirect means such as cardiac MRI scans or measuring the voltage of the tissues. During cardiothoracic surgery, tissue from the left atrium is removed as a part of the procedure. This tissue is normally disposed of, but we would propose to consent patients to collect it to allow it to be analysed. Such analysis would examine the composition of the tissue, including the pattern of scarring, to allow us to gain a greater insight into the mechanisms of AF.

DETAILED DESCRIPTION:
During cardiac surgery, a randomised trial has shown that surgical exclusion of the LAA at the time of cardiac surgery is associated with a 2.2% reduction in ischaemic stroke and systemic embolism. Therefore, surgical exclusion of the LAA, which in the latter study was most commonly achieved by excision, is a well-recognised part of routine surgical practice for patients with AF. During lung resections for malignancies, irrespective of a history of AF, along with the part of the lung being resected, the pulmonary vein and surrounding portion of the left atrium are also removed. These operations therefore provide tissue which is known to be of great importance in promoting and sustaining AF, but which is normally discarded.

In the current study proposal, we will obtain this tissue and analyse it histologically. In the first instance, as a pilot study of up to 10 patients to assess the feasibility of such an analysis. This sample size is informed by our previous basic science studies of cardiac and lung fibrosis and will inform the design of a future full study. We aim to obtain samples from patients in sinus rhythm (thoracic surgical patients) and varying durations of AF (all surgical cases) to encompass tissues with different degrees of fibrosis.

Design of research Up to 10 patients undergoing cardiothoracic surgery at University Hospital Southampton NHS Foundation Trust (UHS) will be recruited. In all cases, the patients would be undergoing surgery where the tissue being studied in the protocol would normally be removed. In the case of thoracic surgical patients, this would be those undergoing lung resections where an ostial pulmonary vein segment will be excised. Here the aim will be to have at least one patient with no history of atrial fibrillation, paroxysmal AF and persistent AF. Cardiac surgical patients included will be those where surgical left atrial exclusion will be performed as part of the procedure, in this case at least one patient with paroxysmal and one with persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent for study
* Male or female subjects between 18 and 100 years of age at the time of consent.
* Thoracic surgical patients either with or without a history of AF undergoing lung resection where an ostial pulmonary vein segment will be excised as part of this resection
* Cardiac surgical patients with a history of AF where surgical LAA exclusion is planned as part of the procedure

Exclusion Criteria:

* Patient unable or unwilling to consent
* Patient not having ostial pulmonary vein or left atrial appendage tissue excised as part of routine clinical care.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac and thoracic surgery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Histological analysis | 1 year
  Immunohistochemistry, in situ hybridisation, electron microscopy, collagen cross-linking
Molecular analysis | 1 year
  genome sequencing, miRNA and RNA sequencing, culture, RT-PCR, flow cytometry and immunocytochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Waqas Ullah, Principal Investigator — University Hospital Southampton NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Undecided
All data will be anonymised.